CLINICAL TRIAL: NCT00206596
Title: Randomized, Stratified, Double-Blind, Placebo-Controlled Phase 2 Study of Steroid-Sparing Properties of Sargramostim (Leukine) Therapy in Patients With Cortico-Dependent Crohn's Disease
Brief Title: Study in Patients With Crohn's Disease Who Are Steroid Dependent, Despite Previous Unsuccessful Attempts to Reduce Steroids Due to Worsening of Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 307501; 91282; Novel 2
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — sargramostim

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Sargramostim (Leukine)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sargramostim (Leukine) — Once daily via subcutaneous injection for up 22 weeks
  Other Names: BAY86-5326
  Arms: Arm 1
Drug: Placebo — Once daily via subcutaneous injection for up 22 weeks
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Leukine to decrease the need for steroid treatment for Crohn's disease.

DETAILED DESCRIPTION:
On 29 May 2009, Bayer began transitioning the sponsorship of this trial to Genzyme. NOTE: This study was originally posted by sponsor Berlex, Inc. Berlex, Inc. was renamed to Bayer HealthCare, Inc.

ELIGIBILITY:
Inclusion Criteria:

* You must have active Crohn's disease at screening and been diagnosed with Crohn's disease within 6 months at screening.
* You must have steroid dependent disease (receiving between 10-40 mgs/day prednisone therapy for greater than 3 months prior to screening and had at least one unsuccessful attempt to reduce cortico-steroids due to worsening of disease).
* You must be able to give yourself an injection of study drug or have another person help you give the injection.
* You must not be pregnant and agree to use birth control if you are a sexually active male or female of childbearing potential.

Exclusion Criteria:

* You may not be taking medications not allowed on this study.
* You may not have had GI surgery or bowel obstruction in the last 6 months.
* You may not have ever taken this drug or drugs of similar type in the past.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2003-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Corticosteroid-free remission | At the end of the study treatment

SECONDARY OUTCOMES:
Steroid-free remission or response to treatment as defined by the protocol | At the end of the study treatment
Quality of Life using Inflammatory Bowel Disease Questionaire, SF 36 and EuroQol-derived visual scale (VAS) | At the end of the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company

REFERENCES:
- [Derived] Valentine JF, Fedorak RN, Feagan B, Fredlund P, Schmitt R, Ni P, Humphries TJ. Steroid-sparing properties of sargramostim in patients with corticosteroid-dependent Crohn's disease: a randomised, double-blind, placebo-controlled, phase 2 study. Gut. 2009 Oct;58(10):1354-62. doi: 10.1136/gut.2008.165738. Epub 2009 Jun 7. PMID 19505878